CLINICAL TRIAL: NCT00445562
Title: Breast Cancer Siblings Database
Brief Title: Blood Sample Collection and Health Information Collection From Patients With Invasive Breast Cancer and Their Brothers and Sisters
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: GenBasix Incorporated (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: GENBASIX-00127; CDR0000529353 (Registry Identifier: PDQ (Physician Data Query)); GENBASIX-1024122
Record Dates: First submitted 2007-03-07; First posted 2007-03-09 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2009-07

CONDITIONS: Breast Cancer
Keywords: male breast cancer; recurrent breast cancer; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male

INTERVENTIONS:
Other: biologic sample preservation procedure
Other: informational intervention

SUMMARY:
RATIONALE: Collecting blood samples and health information from patients with invasive breast cancer and from their brothers and sisters over time may help the study of cancer in the future.

PURPOSE: This study is collecting blood samples and health information over time from patients with invasive breast cancer and from their brothers and sisters.

DETAILED DESCRIPTION:
OBJECTIVES:

* Collect blood samples and medical and background information from patients with invasive breast cancer and their affected or unaffected siblings.

OUTLINE: Patients and their siblings undergo blood collection. They also complete medical and background questionnaires.

Patients and their siblings are followed annually for 5 years.

PROJECTED ACCRUAL: A total of 1,000 patients and siblings will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Pathologically confirmed invasive breast cancer (patient)

    * No ductal carcinoma in situ
  * Affected OR unaffected sibling

    * Affected sibling must have had (or currently has) breast cancer only
    * Unaffected sibling must be female
    * No deceased siblings
    * Must be a full-blood related sibling
* Patients receiving treatment on clinical trial ECOG-E1Y97 or ECOG-E3Y92 are not eligible

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2001-01; Primary Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Collection of blood samples and medical and background information

CONTACTS AND LOCATIONS:
Overall Officials: Richard A. Shapiro, MD, Study Chair — GenBasix Incorporated
Locations (1):
- GenBasix Incorporated, Duarte, California, United States